CLINICAL TRIAL: NCT00727077
Title: Treatment of Chronic Hepatitis C in Children With Intron Vial or Pen and Rebetol According to German Law (§ 67 Abs 6 AMG)
Brief Title: Post-marketing Surveillance of Children With Chronic Hepatitis C Treated With Intron A (Vial or Pen) and Rebetol (Study P04397)(TERMINATED)
Status: Terminated | Type: Observational
Why Stopped: Study halted due to low recruitment. The 3 participants at time of termination transferred into study P04538 (NCT00727077). See NCT00727077 for details/results.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04397
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Interferon alpha-2; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IntronA/Rebetol: Children age 3 to 17, with chronic hepatitis C, treated in clinical practice at 10 German sites
  Interventions: Biological: IntronA (interferon alfa-2b; SCH 30500); Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: IntronA (interferon alfa-2b; SCH 30500) — IntronA (3 Mio I.E./m2, 3 times per week) administered in accordance with the SPC and approved European labeling
  Other Names: SCH 30500
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol (15 mg/kg/day) administered in accordance with the SPC and approved European labeling
  Other Names: SCH 18908

SUMMARY:
The objective of the study is to assess the safety and efficacy of Intron A (3 Mio I.E./m2, 3 times per week) and Rebetol (15 mg/kg/day) in children aged 3 to 17, treated in common medical practice at 10 sites in Germany. The primary objective is to determine if there are any new severe adverse events observed with this recently approved dosing regimen. The study will also evaluate the rates of eradication of the HCV virus.

This study was terminated due to low enrollment. At the time of termination, 3 participants had enrolled. Therefore, these 3 participants transferred into study P04538 (NCT00727077) and will be included in the P04538 (NCT00727077) data reporting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C (serum HCV-RNA-positive)
* Age 3 to 17 years
* Treatment-naïve
* Platelets >= 100,000/mm^3
* Neutrophil counts >= 1,500/ mm^3
* TSH must be within normal limits
* Hemoglobin >=12 g/dL (females); >=13 g/dL (males)
* Women of childbearing potential must have a routine pregnancy test performed monthly during treatment and for 7 months thereafter. Sexually active female subjects of childbearing potential must be practicing adequate contraception (intrauterine device, oral contraceptives, implanted contraceptives, surgical sterilization, barrier method, or monogamous relationship with a male partner who has had a vasectomy or is using a condom (+ spermicide) during the treatment period and for 7 months after stopping treatment.
* Sexually active male subjects must be practicing acceptable methods of contraception (vasectomy, use of condom + spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 7 months after stopping treatment.

Exclusion Criteria:

* Contraindications according to the SPC and European approval
* Pretreatment of chronic hepatitis C
* Liver decompensation
* Hypersensitivity to the active substance or to any interferons or to any of the excipients
* Pregnant woman
* Woman who are breast feeding
* Existence of or history of psychiatric condition, in particular depression, suicidal ideation or suicide attempt
* A history of severe pre-existing cardiac disease, including unstable or uncontrolled cardiac disease in the previous six months
* Severe debilitating medical conditions, including patients with chronic renal failure or creatinine clearance < 50 mlLmin
* Autoimmune hepatitis or history of autoimmune disease
* Severe hepatic dysfunction or decompensated cirrhosis of the liver
* Pre- existing thyroid disease unless it can be controlled with conventional therapy
* Epilepsy and/or compromised central nervous system function
* Individual decision of physician if patient suitable for treatment (e.g., disturbance of growth)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children age 3 to 17 years, with chronic hepatitis C, treated in clinical practice at 10 German sites
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events | After the inclusion of the subject in the study (defined as the time when the subject signs the informed consent) and up to 30 days after the subject completed or discontinued the study

SECONDARY OUTCOMES:
Sustained virologic response (defined as undetectable viral load at 24 weeks post-treatment) | Assessed at the end of treatment and 24 weeks post-treatment